CLINICAL TRIAL: NCT06102265
Title: Effect Of Reusing the Operative Supplies On Cataract Surgery and Climate Change
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hany Mahmoud,MD, ophthalmology lecturer, Sohag University
Other Study IDs: soh-med-23-10-06PD
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Ophthalmopathy
MeSH Terms: conditions — Eye Diseases | interventions — Sterilization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1: In one arm of the study group, the surgeon changed the gown and the glove between each case with hand sterilization with alcohol before and after wearing the next glove.
  Each keratome and MVR were used for multiple patients until they became blunt. We used the same IOL cartridge for every three cases and the same OVD in multiple patients. We immersed keratome, MVR, IOL cartridge, and cannulas of OVD in alcohol between cases.
  As regard the phaco machine, we used Alcon Infiniti and Alcon Centurion and the same tip for all cases. The tip was immersed in a test chamber filled with alcohol between cases and not changed until we noticed a morphological change or they became blunt. Also, the same cassette was used in multiple surgeries and changed after collecting the plastic bag full of fluid.
  Interventions: Procedure: sterilization
- group 2: In another arm, we used the same steps except that the surgeon changed the glove only and used alcohol for hand sterilization before and after wearing the next glove. One gown was used for all the cases. As regard the intracameral antibiotic prophylaxis, a bottle of Vigamox, 5ml, was withdrawn, and each 1 ml was diluted with 5 ml saline. Using this dilution, 0.1 ml was injected intracamerally at the end of the operation. Finally, we did corneal hydration of the main wound and the side ports.
  Interventions: Procedure: sterilization

INTERVENTIONS:
Procedure: sterilization — the use of sterilization methods and the reuse of gowns

SUMMARY:
Although postoperative infectious endophthalmitis and toxic anterior segment syndrome (TASS) rarely happen, they can threaten sight and are considered complications of intraocular and cataract surgery1.

Reusing surgical supplies during cataract surgery, especially in developing countries, will have a treble impact in lowering the financial costs of surgery, the emissions of greenhouse gas, and environmental waste. Nearly half the waste of cataract surgery is recyclable, as reported by a prospective Malaysian study 8.

Despite the increasing evidence of reusing the operative supplies, numerous healthcare professionals may be reluctant to consider it due to worries about cross-contamination among patients2.

According to the Aravind Eye Care System (AECS) in Tamil Nadu, India, endophthalmitis rated 0.02% in over a million consecutive cataract cases despite the observation that cannulas, irrigation/ aspiration tubing, gowns, surgical gloves, irrigating bottles, as well as topical and intraocular drugs are normally recycled to cut cost and waste3,4.

On the other hand, health care plays a key role in climate change, as well as financial and environmental waste2. Cataracts are the leading cause of blindness and visual impairment worldwide, making cataract surgery one of the most performed surgical procedures5. The carbon footprint of cataract surgery, especially phacoemulsification, is a significant research field6-8.

In the United Kingdom, cataract surgery releases 180 kg of CO2- equivalents per eye, causing over half of the emissions due to obtaining large disposable medical equipment9. In ACES, phacoemulsification generated 5.9 kg of carbon emissions4.

In comparison to the United Kingdom and the United States of America, the cataract surgery's low rates of infection in AECS were accomplished with 1/10 supply costs and 1/20 global warming emissions6.

Being the most performed operation, cataract surgery and ophthalmology, in general, can meaningfully influence lowering environmental and economic waste in their surgical services1.

The aim of this work is to show if reusing the operative supplies to reduce financial costs, especially in developing countries, and to lower global warming and climate change will affect the rate of postoperative endophthalmitis after cataract surgery

DETAILED DESCRIPTION:
Although postoperative infectious endophthalmitis and toxic anterior segment syndrome (TASS) rarely happen, they can threaten sight and are considered complications of intraocular and cataract surgery1.

Reusing surgical supplies during cataract surgery, especially in developing countries, will have a treble impact in lowering the financial costs of surgery, the emissions of greenhouse gas, and environmental waste. Nearly half the waste of cataract surgery is recyclable, as reported by a prospective Malaysian study 8.

Despite the increasing evidence of reusing the operative supplies, numerous healthcare professionals may be reluctant to consider it due to worries about cross-contamination among patients2.

According to the Aravind Eye Care System (AECS) in Tamil Nadu, India, endophthalmitis rated 0.02% in over a million consecutive cataract cases despite the observation that cannulas, irrigation/ aspiration tubing, gowns, surgical gloves, irrigating bottles, as well as topical and intraocular drugs are normally recycled to cut cost and waste3,4.

On the other hand, health care plays a key role in climate change, as well as financial and environmental waste2. Cataracts are the leading cause of blindness and visual impairment worldwide, making cataract surgery one of the most performed surgical procedures5. The carbon footprint of cataract surgery, especially phacoemulsification, is a significant research field6-8.

In the United Kingdom, cataract surgery releases 180 kg of CO2- equivalents per eye, causing over half of the emissions due to obtaining large disposable medical equipment9. In ACES, phacoemulsification generated 5.9 kg of carbon emissions4.

In comparison to the United Kingdom and the United States of America, the cataract surgery's low rates of infection in AECS were accomplished with 1/10 supply costs and 1/20 global warming emissions6.

Being the most performed operation, cataract surgery and ophthalmology, in general, can meaningfully influence lowering environmental and economic waste in their surgical services1.

The aim of this work is to show if reusing the operative supplies to reduce financial costs, especially in developing countries, and to lower global warming and climate change will affect the rate of postoperative endophthalmitis after cataract surgery Preoperatively, all patients underwent routine systemic examinations, such as blood pressure and blood glucose level measurements, ECG, and hepatitis markers.

No preoperative topical antibiotics prophylaxis was described for all patients. Retrobulbar and peribulbar anesthesia were used for all patients. While performing the anesthesia, a drop of topical anesthesia, a drop of povidone-iodine 5%, and a drop of Moxifloxacin (Vigamox) were installed in the conjunctival cul-de-sac immediately prior to the surgery. Topical povidone-iodine was utilized immediately prior to the surgery in order to prepare the periorbital area (10%). After opening the face drape, a drop of povidone-iodine 5% was also installed in the conjunctival sac and washed thoroughly before starting the operation.

Topical Gatifloxacin (Tymer) and Prednisolone (Optipred)drops were instilled four times daily in the first 10 days following the surgery. Additionally, a topical combination solution of Ofloxacin, dexamethasone (Dexaflox), and a lubricant(Systane) was used three times daily for the next four weeks.

Hand sterilization of the surgeon and the assistant was done once before starting the first case with povidone-iodine and alcohol.

In one arm of the study group, the surgeon changed the gown and the glove between each case with hand sterilization with alcohol before and after wearing the next glove.

Each keratome and MVR were used for multiple patients until they became blunt. We used the same IOL cartridge for every three cases and the same OVD in multiple patients. We immersed keratome, MVR, IOL cartridge, and cannulas of OVD in alcohol between cases.

As regard the phaco machine, we used Alcon Infiniti and Alcon Centurion and the same tip for all cases. The tip was immersed in a test chamber filled with alcohol between cases and not changed until we noticed a morphological change or they became blunt. Also, the same cassette was used in multiple surgeries and changed after collecting the plastic bag full of fluid.

We routinely used intracameral Moxifloxacin (Vigamox) as antibiotic prophylaxis. The bottle of 5ml was withdrawn, put in the irrigating bottle of phacoemulsification, used throughout the operation, and used for multiple patients until the bottle became empty.

In another arm, we used the same steps except that the surgeon changed the glove only and used alcohol for hand sterilization before and after wearing the next glove. One gown was used for all the cases. As regard the intracameral antibiotic prophylaxis, a bottle of Vigamox, 5ml, was withdrawn, and each 1 ml was diluted with 5 ml saline. Using this dilution, 0.1 ml was injected intracamerally at the end of the operation. Finally, we did corneal hydration of the main wound and the side ports.

ELIGIBILITY:
Inclusion Criteria:

* adults with cataract not diabetics not hypertensive

Exclusion Criteria:

youngs diabetics hypertensive

-

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with cataract subjected to phcoemulsification
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
postoperative complications | 6 months
  rate of occurence of infection

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Sohag University, Sohag
  - Hany Mahmoud, Sohag

IPD SHARING:
Plan to Share IPD: Undecided